CLINICAL TRIAL: NCT07240597
Title: Acute Effects of Different Potentiation Protocols During Warm-Up in Competitive Young Swimmers: A Randomized Crossover Trial
Brief Title: Acute Effects of Different Warm-Up Protocols in Competitive Young Swimmers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Giacomo Belmonte, Dr., University of Palermo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 62141-2025-2; 311/2025 (Other: Bioethics Committee- University of Palermo)
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Athletes; Post Activation Potentiation; Countermovement Jump; Performance; Warm-up

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Band Squats (BS) (Experimental): The band squats protocol consists of four sets of four repetitions with two minutes of recovery between sets. Four elastic bands of different resistance will be tested for each participant, and the correct band will be used. During the protocol, subjects will stop at the same depth as a swimming start, with a knee angle between 135 and 145°. All subjects will receive verbal encouragement during the performance in the same way.
  Interventions: Other: Squats with resistance band
- Drop Jump (DJ) (Experimental): The drop jump protocol consists of three sets of five repetitions of jumping after falling from a 45 cm box, with a fifteen-second break to reposition over the box and three minutes of recovery between sets.
  Interventions: Other: Vertical jump after dropping from a box
- Band Squats (BS) + Drop Jump (DJ) (Experimental): A combination of the band squats and the drop jumps
  Interventions: Other: Combination BS + DJ
- Control Group (CG) (No Intervention): Control Group

INTERVENTIONS:
Other: Squats with resistance band — The elastic band squat protocol consisted of four sets of four repetitions with two minutes of recovery between sets (estimated total time: 9 minutes). Participants in a standing position should take one of the four elastic resistance bands (GymBeam), anchor it under their feet, and under each shoulder.
  Arms: Band Squats (BS)
Other: Vertical jump after dropping from a box — A box for plyometric training (Yes4All) will be used in its 45 cm height section. The protocol consists of three sets of four repetitions. Fifteen seconds of recovery time will be allowed to reposition above the box, and three minutes of recovery time between sets (estimated total time: 10 minutes). Participants will be encouraged to reach maximum height with each jump, without bending their knees during the flight phase.
  Arms: Drop Jump (DJ)
Other: Combination BS + DJ — A combination of squats with an elastic band and vertical plyometric jump after dropping from a box. The protocols are the same as those described in the other interventions (total estimated time: 19 minutes).
  Arms: Band Squats (BS) + Drop Jump (DJ)

SUMMARY:
Several warm-up strategies are commonly employed by athletes to optimize athletic performance and minimize the risk of injury. Recently, Post-Activation Performance Enhancement (PAPE) has been demonstrated to be effective in improving athletic performance. Nevertheless, the difference with the general warm-up is still unclear and poorly studied. Conventionally, short-term performance improvements achieved after brief periods of maximal activity have been attributed to PAP, a muscle memory mechanism that generates involuntary and short-lived effects (~28 seconds). This condition appears to be activated only by a history of localized maximal contractions. In the literature, various conditioning protocols with differing durations and intensities have been explored, often finding conflicting results in terms of athletic performance. In swimming, few PAPE warm-up protocols outside the pool have been studied, despite their potential usefulness considering the waiting times before competitions.

Therefore, this study explores the effects of three different warm-up protocols in young swimmers. Specifically, different exercise protocols will be included in the athletes' usual warm-up routine, aimed at improving athletic performance through PAPE effects. In line with existing literature, the performance parameters examined are the countermovement jump (CMJ) and the times recorded for covering race distances ( 25 m, 50 m, 100 m). In addition, skin temperature, heart rate (HR), muscle oxygen saturation (SmO2), and perceived exertion (RPE) are also measured after the protocols to investigate possible relationships with performance measures. Nevertheless, the primary aim of this study is to compare different warm-up protocols in young swimmers to maximize their athletic performance.

DETAILED DESCRIPTION:
All outcome data will be expressed as mean ± standard deviation. The first warm-up section for all athletes will take place in the pool. Subsequently, baseline assessments (T0) will be conducted. Through a randomized study design, each participant will perform three plyometric protocols (squats with elastic bands, box jumps, or a combination of both).

To examine differences in the main outcomes, a repeated-measures ANOVA (4 conditions x 5 time points) will be conducted. When a significant condition × time interaction is detected, post hoc analyses to determine specific between and within-group differences. Effect sizes will be reported as partial eta squared (η²p). Statistical significance will be set at p < 0.05 for all analyses

ELIGIBILITY:
Inclusion Criteria:

* Active participation in competitive training programs (at least 10 hours per week), at least one year of experience in competitions organized by the Italian Swimming Federation, and no recent injuries.
* Experience of resistance training for at least 6 months

Exclusion Criteria:

* Irregular training participation
* History of injuries in the 6 months prior to the study

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Counter Movement Jump (CMJ) | Before the start of the investigated warm-up phase (baseline, T0), 15 seconds after the protocols (T1), 3 minutes after the protocols (T2), 6 minutes after the protocols (T3), 9 minutes after the protocols (T4), 12 minutes after the protocols (T5)
  Initially, the athlete stands upright on a flat surface or force platform, feet shoulder-width apart, hands on hips (to eliminate arm swing). Without a pause, the athlete performs a quick downward movement (countermovement) by bending the knees and hips, then immediately jumps vertically as high as possible. The athlete lands in an upright position on the same spot, trying to absorb the impact with knees slightly bent. Jump height and flight time is recorded using an optical system, Optojump™ system(Microgate, Bolzano, Italy) connected to a personal computer with dedicated software(OptojumpTM Next software). The system consists of two optical bars, a receiver and a transmitter, positioned 1m apart. The bars identify ground contact time(with a precision of 1ms) and then convert non-contact time into cm. Based on recommendations on optimal jump height (20 to 60cm).
Time Swimming Trials | Before the start of the investigated warm-up phase (baseline, T0) and after the individual time of recovery resulting from the height of the CMJ (T1)
  In a second moment, after establishing the best warm-up protocol (from among those proposed) with the best recovery (derived from the CMJ height with the time ratio) for each individual, the 25, 50, and 100 m measurements will be evaluated in the pool. This will take place at a later stage in a 25 m pool. The first part of the warm-up will be the same for all subjects, while the second part will be personalized, based on their Post Activation Performance Enhancement.

SECONDARY OUTCOMES:
Skin Temperature | Before the start of the investigated warm-up phase (baseline, T0), 15 seconds after the protocols (T1), 3 minutes after the protocols (T2), 6 minutes after the protocols (T3), 9 minutes after the protocols (T4), 12 minutes after the protocols (T5)
  The FLIR Foedge thermal imaging camera will be used to capture high-resolution thermal images of the target muscle area under controlled environmental conditions. The thermal imaging camera will be positioned approximately 0.5 meters from the subject's skin surface, with a fixed focal length lens to ensure sharp images. The room will be continuously monitored for temperature and humidity, minimizing external thermal influences. Ambient lighting will be kept low to avoid thermal interference from light sources. The thermal imaging camera will be calibrated before each session, connected to the same smartphone, and images will be captured at a frequency of 30 Hz to monitor temperature changes in real-time before and after muscle activity.
Heart Rate (HR) | Before the start of the investigated warm-up phase (baseline, T0), 15 seconds after the protocols (T1), 3 minutes after the protocols (T2), 6 minutes after the protocols (T3), 9 minutes after the protocols (T4), 12 minutes after the protocols (T5)
  Heart rate (HR) will be measured with a Polar H10 chest strap sensor, a device known to give accurate results. To prepare, participants were asked not to drink coffee or alcohol, avoid hard exercise for 24 hours, and keep their normal sleep routine. The tests will always be done at the same time of day in every condition to avoid daily rhythm effects. The average HR over two minutes of recording will be recorded. The chest strap will be placed just below the chest bone and secured around the chest. Once the signal was ready, data will sent automatically to a mobile app (Elite HRV). All data will be later analyzed with special software (Kubios HRV).
Muscle Oxygen Saturation (SmO2) | Before the start of the investigated warm-up phase (baseline, T0), 15 seconds after the protocols (T1), 3 minutes after the protocols (T2), 6 minutes after the protocols (T3), 9 minutes after the protocols (T4), 12 minutes after the protocols (T5)
  The Moxy oxygen sensor will be positioned on the vastus lateralis portion of the quadriceps muscle to monitor muscle oxygenation dynamics before, during and after exercise. The probe will be securely attached using the appropriate elastic band to minimize motion artifact and oriented parallel to the muscle fibers. Data acquisition will performed at a sampling rate of 10 Hz, capturing relative changes in muscle oxygen saturation (SmO2) and total hemoglobin concentration. The site will be carefully cleaned and shaved when necessary to ensure optimal sensor contact. This setup allows for real-time, non-invasive assessment of local muscle oxygen utilization and hemodynamics, which is useful for evaluating muscular fatigue and metabolic responses.
Ratings of perceived exertion (RPE) | Before the start of the investigated warm-up phase (baseline, T0), 15 seconds after the protocols (T1), 3 minutes after the protocols (T2), 6 minutes after the protocols (T3), 9 minutes after the protocols (T4), 12 minutes after the protocols (T5)
  The Rate of Perceived Exertion (RPE) scale will be employed to assess participants' subjective perception of exercise intensity during the protocol. The Borg Scale will be used following the pool warm-up, before each testing session, after each testing session, and at study conclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- A.S.D. Swim Power, Bagheria, Palermo, Italy